CLINICAL TRIAL: NCT06677086
Title: Effect of HIFEM Application on Musculoskeletal System: Evaluation of Musculoskeletal System Improvement
Brief Title: HIFEM for Musculoskeletal System Improvement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: BTL Industries Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BTL-899_CTUS900
Record Dates: First submitted 2024-11-05; First posted 2024-11-06 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2024-12

CONDITIONS: Muscle Disorder; Musculoskeletal Diseases
Keywords: muscle; musculoskeletal system; extremities
MeSH Terms: conditions — Muscular Diseases; Musculoskeletal Diseases | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Treatment with BTL-899 (Experimental): Four (4) BTL-899 treatments will be applied to the impaired musculoskeletal area, either on the upper or lower extremity.
  Interventions: Device: Treatment with BTL-899

INTERVENTIONS:
Device: Treatment with BTL-899 — The treatment administration phase will consist of four (4) treatments, delivered 5-10 days apart. The applicators of BTL-899 device will be applied over the designated area. Each treatment session will last 30 minutes.

SUMMARY:
The goal of this clinical trial is to investigate the effect of the BTL-899 device on improving the Musculoskeletal System in healthy adult volunteers. The main question it aims to answer is:

Whether the BTL-899 device is able to change musculoskeletal system perception before and after treatment, based on the Subject Satisfaction questionnaire.

Participants will complete four treatments, and two follow-up visits.

DETAILED DESCRIPTION:
This study will evaluate the clinical efficacy and performance of the BTL-899 device for changes in the musculoskeletal system, specifically of the upper and lower extremities. The study is a prospective, multi-center, open-label, single-arm study. The subjects will be enrolled and assigned into a single study group. Subjects will be required to complete four (4) treatment visits and two follow-up visits. All of the study subjects will receive the treatment with the study device.

At the baseline visit, the subject's weight will be recorded and subjects will fill in the Western Ontario and McMaster Universities questionnaire.

The treatment administration phase will consist of four (4) treatments, delivered 5-10 days apart. The applicators of BTL-899 will be applied over the designated area. Each therapy session will last 30 minutes.

At the last therapy visit, the subject's weight will be recorded. In addition, subjects will receive Therapy Comfort, Subject Satisfaction Questionnaire and Western Ontario and McMaster Universities questionnaire to fill in.

Safety measures will include documentation of adverse events (AE), which will be assessed after each procedure and at all of the follow-up visits.

During the post-procedure visits (at 1-month and 3-month follow-up visits), the subject's satisfaction, Western Ontario and McMaster Universities questionnaire, and weight will be recorded. In addition, subjects will receive a Lifestyle Change Questionnaire to fill in.

ELIGIBILITY:
Inclusion Criteria:

* Age 22 years and older
* Voluntarily signed an informed consent form
* BMI ≤ 35 kg/m2
* Women of child-bearing potential* are required to use birth control measures during the whole duration of the study
* Subjects willing and able to abstain from partaking in any treatments other than the pre-procedure therapy regime and the study procedure for improvement of the musculoskeletal system
* Subjects willing and able to maintain their regular (pre-procedure) diet, exercise and therapy regimen without affecting significant change in either direction during study participation

Exclusion Criteria:

* Electronic implants (such as cardiac pacemakers, defibrillators, and neurostimulators)
* Metal implants
* Drug pumps
* Malignant tumor
* Pulmonary insufficiency
* Application over muscles in acute phase of injury
* Cardiovascular diseases
* Disturbance of temperature or pain perception
* Hemorrhagic conditions, blood coagulation disorders or anticoagulation therapy.
* Septic conditions and empyema
* Acute inflammations
* Systemic or local infection such as osteomyelitis and tuberculosis
* Contagious skin disease
* Elevated body temperature
* Pregnancy, postpartum period, nursing, and menstruation
* A metal-containing intrauterine device (IUD)
* Graves' disease

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2024-05-08 (Actual); Primary Completion 2025-01-22 (Actual); Study Completion 2025-01-22 (Actual)

PRIMARY OUTCOMES:
Musculoskeletal System Perception | 15 months
  The evaluation of changes in musculoskeletal system perception before and after treatment will be based on the 5-point Likert Scale Subject Satisfaction questionnaire. Responses to questions about the treated musculoskeletal area will range from "strongly agree" (1 point) to "strongly disagree" (5 points). A higher score for each statement indicate better outcomes. The Subject Satisfaction Questionnaire will be administered after the final treatment, as well as at the 1-month and 3-month follow-up visits.

SECONDARY OUTCOMES:
Incidence of Treatment-related Adverse Events | 15 months
  To evaluate the safety of the device and determine side effects and adverse events (AE) associated with the BTL-899 treatment of the musculoskeletal system through monitoring of adverse reactions and side effects.
Comfort Assessed by Therapy Comfort Questionnaire | 15 months
  Therapy Comfort questionnaire will be used for evaluating the comfort during the treatment sessions. Therapy Comfort questionnaire consists of the question "I found the treatment comfortable", to which responses are based on a 5-point Likert scale (1 = "strongly disagree", and 5 = "strongly agree") and the 10-point Numeric Pain Rating Scale (0 = no pain, 10 = worst possible pain"). A higher score for the statement "I found the treatment comfortable", and lower score on the Numeric Pain Rating Scale indicate higher therapy comfort. The Therapy Comfort questionnaire will be given to subjects after the last treatment.
Physical Function Assessed by the Western Ontario and McMaster Universities questionnaire. | 15 months
  Changes in physical function post-treatment will be assessed using the Western Ontario and McMaster Universities (WOMAC) questionnaire. This 24-item questionnaire measures five items for pain (score range 0-20), two for stiffness (score range 0-8), and 17 for functional limitation (score range 0-68). Improvement is considered a decrease in the obtained score. The questionnaire will be administered at the baseline visit, after the final treatment, and during both follow-up visits at 1 month and 3 months post-treatment.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Trokhan Orthopaedics LLC, Closter, New Jersey
  - New York Orthopedic Hand Surgery, Brooklyn, New York
  - Southeast Texas Orthopedic Group, Houston, Texas